CLINICAL TRIAL: NCT05528367
Title: Tirelizumab in Combination With Chemoradiation in Patients With Unresectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma：A Single Arm Phase II Clinical Study
Brief Title: Tirelizumab in Combination With Chemoradiation in Patients With Unresectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Liu luying, Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZhejiangCH20211029
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2021-10

CONDITIONS: Locally Advanced Gastric Cancer
Keywords: chemoradiotherapy; tirelizumab
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CRT with Tirelizumab (Experimental): Chemotherapy+Tirelizumab:PS regimen:S-1:BSA <=1.25 m2 ,80 mg daily; 1.25 m2 <BSA <1.5 m2,100 mg daily; BSA>=1.5 m2 ,120 mg daily.
  Nab-PTX:preoperation：130mg/m2,d1，8，q3w；adjuvant:100mg/m2,d1，8，q3w； Tirelizumab：200mg d1 q3w.
  Concurrent Chemoradiotherapy:
  Radiation: 45-50Gy/25Fx;During radiation: Nab-PTX:100mg qw,Tirelizumab：200mg d1 q3w.
  Chemotherapy+Tirelizumab:PS regimen:S-1:BSA <=1.25 m2 ,80 mg daily; 1.25 m2 <BSA <1.5 m2,100 mg daily; BSA>=1.5 m2 ,120 mg daily.
  Nab-PTX:preoperation：130mg/m2,d1，8，q3w； Tirelizumab：200mg d1 q3w.
  We will evaluate whether the tumor could be resectable through CT scan and Endoscope after two cycles of Chemotherapy+Tirelizumab and CRT.If it could be resctable,three cycles of adjuvant chemotherapy+Tirelizumab will be arranged;If not,another three cycles of chemotherapy+Tirelizumab will be arranged，then evaluate again.
  Interventions: Drug: Nab-PTX,S-1,Tirelizumab; Radiation: Chemoradiation

INTERVENTIONS:
Drug: Nab-PTX,S-1,Tirelizumab — S-1:BSA <=1.25 m2 ,80 mg daily; 1.25 m2 <BSA <1.5 m2,100 mg daily; BSA>=1.5 m2 ,120 mg daily.
  Nab-PTX:130mg/m2,d1，8，q3w；100mg qw(during radiation) Tirelizumab：200mg d1 q3w.
Radiation: Chemoradiation — 45-50Gy/25F

SUMMARY:
To evaluate the efficacy and safety of chemoradiotherapy combined with tirelizumab in the treatment of initial unresectable locally advanced gastric cancer or gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged ≥ 18 years; ≤ 75 years old;
2. The histopathology confirmed the diagnosis of previously untreated locally advanced unresectable HER2 negative gastric or gastroesophageal junction adenocarcinoma (imaging evaluation showed that the primary tumor was severely invaded, could not be separated from the surrounding normal tissue, or had surrounded large blood vessels, or regional lymph nodes were fixed and fused, or the metastatic lymph nodes were not within the scope of surgical clearance), and there was no peritoneal metastasis during laparoscopic exploration;
3. There is no serious liver and kidney function damage, and the functional level of organs must meet the following requirements: ANC ≥ 1.5 × 109/L； PLT ≥ 90 × 109/L； Hb ≥ 90 g/L； TBIL ≤ 1 × ULN； ALT and AST ≤ 1.5 × ULN，ALP ≤ 2.5 × ULN； Bun and Cr ≤ 1 × ULN and creatinine clearance ≥ 50 ml / min (Cockcroft Gault formula); LVEF ≥ 50%； The QT interval (QTCF) corrected by fridericia method was < 450 ms in males and < 470 MS in females; INR ≤ 1.5 × ULN，APTT ≤ 1.5 × ULN；
4. The patient has at least one measurable lesion, which is evaluated by the investigator according to (RECIST) v1.1;
5. ECoG PS score 0 or 1;
6. Life expectancy ≥ 6 months;
7. The investigator assessed that the patient could comply with the protocol requirements;
8. Sign the informed consent document.

Exclusion Criteria:

1. Received systemic cytotoxic drug chemotherapy;
2. Patients with hypersensitivity or hypersensitivity to therapeutic drugs and patients with autoimmune diseases; Have received allogeneic tissue / solid organ transplantation;
3. There is third space effusion (such as pleural fluid and ascites) that cannot be controlled by drainage or other methods;
4. Use steroids for more than 50 days, or need to use steroids for a long time;
5. Uncontrolled symptomatic brain metastases or mental disorders cannot correctly express subjective symptoms;
6. The abnormal coagulation function has clinical significance, has bleeding tendency or is receiving thrombolytic or anticoagulant treatment;
7. Unable to swallow, chronic diarrhea and intestinal obstruction, and there are many factors affecting drug taking and absorption;
8. Other malignant tumors occurred within 5 years before enrollment, except for cervical carcinoma in situ or skin squamous or basal cell carcinoma that had been treated for radical cure before;
9. Pregnant or lactating women who have fertility but refuse to take contraceptive measures;
10. Those with serious heart disease or medical history, including: recorded history of congestive heart failure, high-risk uncontrollable arrhythmia, angina pectoris requiring medical treatment, clinically clear heart valve disease, history of serious myocardial infarction and stubborn hypertension;
11. According to the judgment of the investigator, there are concomitant diseases (such as uncontrolled hypertension, diabetes, thyroid disease, etc.) that seriously endanger the patient's safety or affect the patient's completion of the study;
12. The investigator determines that other conditions are not suitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of resectable patients with negative incisal margin R0 resection rate | 18 weeks after treatment completion
  the rate of resectable patients with negative incisal margin

CONTACTS AND LOCATIONS:
Locations (1):
- Liu luying, Hangzhou, Zhejiang, China